CLINICAL TRIAL: NCT01226043
Title: An Open Label Randomized Multicenter Study to Assess Patient Preference for and Evaluate Clinical Benefit of Insulin Glargine (Lantus®) SoloSTAR® Pen Versus Conventional Vial/Syringe Method of Insulin Glargine (Lantus®) Injection Therapy in Patients With Type 2 Diabetes Mellitus
Brief Title: Patient Preference and Satisfaction With Insulin Glargine (Lantus) Solostar Pen vs Conventional Vial-Syringe Method of Lantus Injection Therapy in Patients With Type 2 Diabetes Mellitus
Acronym: Pen Preference
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_05191; U1111-1116-3054 (Other: UTN)
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (2):
- Lantus (insulin glargine) vial & syringe (Experimental): 10 mL vial, 1000 U per vial for subcutaneous administration once a day. Starting dose will be 0.2 Unit per kilogram of body weight.
  Interventions: Drug: Insulin Glargine
- Lantus (insulin glargine) SoloSTAR pen (Experimental): 3 mL SoloSTAR pre-filled disposable insulin delivery device (pen), 300 U per device for subcutaneous administration once a day. Starting dose will be 0.2 Unit per kilogram of body weight.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — * Pharmaceutical form: solution for injection
  * Route of administration: subcutaneous
  Other Names: Lantus

SUMMARY:
Primary Objective:

To assess patient preference for Lantus SoloSTAR pen versus Lantus vial and syringe at the end of Crossover Phase (Week 4) in patients with type 2 diabetes mellitus (T2DM)

Secondary Objectives:

To compare Lantus SoloSTAR pen versus Lantus vial and syringe with regard to the following parameters:

Randomization/Crossover phase:

* Healthcare professional's (HCP) recommendation for Lantus SoloSTAR pen versus Lantus vial and syringe

Re-randomization phase:

* Change in Fasting Plasma Glucose (FPG) from week 4 to week 10
* Percentage of patients achieving FPG<110 mg/dL at week 10
* Change in Lantus dose injected per day (U) from week 4 to week 10

Observational phase:

* Percentage of patients achieving glycosylated hemoglobin (HbA1c) goal (<7%) at week 40
* Time to first observation of HbA1c<7% during the observational phase
* Percentage of patients who discontinue Investigational Product (IP) during the observational phase due to dissatisfaction with their current device

All phases:

* Percentage of patients who discontinue IP during each phase of the study
* Safety assessment such as occurrence of hypoglycemic events (HE) and adverse events (AE)

DETAILED DESCRIPTION:
This study consisted of a 1 week Screening Phase, a 4-week Randomization/Crossover Phase, a 6-week Re-randomization Phase, followed by a 30 week Observational Phase.

The total duration of study participation was up to 41 weeks with a total treatment duration of up to 40 weeks of Lantus exposure.

ELIGIBILITY:
Inclusion criteria:

Patients with a confirmed diagnosis of type 2 diabetes mellitus who were treated with any combination of 2 or 3 oral antidiabetic drugs (OADs) at a stable dose for the preceding 3 months, including but not limited to:

* Metformin + sulfonylurea + thiazolidinedione (Pioglitazone)
* Metformin + sulfonylurea
* Metformin + thiazolidinedione (Pioglitazone)
* Metformin + dipeptidyl peptidase (DPPIV)

And for whom the Investigator/treating physician had decided that basal insulin was appropriate.

Patients who had signed an Informed Consent Form and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form

Exclusion criteria:

* Patients less than 18 years or greater than 85 years of age (ie, have not reached the age of 86 at the screening visit)
* Patients with a confirmed diagnosis of type 1 diabetes mellitus
* Patients who were treated with insulin or who had been treated with insulin in the preceding 12 months with the exception of insulin treatment during hospitalization (ie, patients who received insulin while hospitalized could be included)
* Patients whose screening HbA1c is <7% or >10%
* Patients with current addiction or current alcohol / drug abuse
* Patients with cardiac status New York Heart Association III-IV
* Patients with stroke, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, or unstable angina pectoris within the 12 months prior to screening
* Patients with a diagnosis of dementia, severe visual or dexterity impairment
* Patients with any malignancy within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or adequately treated cervical carcinoma in situ
* Patients with concomitant disease or concomitant medication that could interfere with treatment or ability to answer questionnaires
* Patients who were unable to self-inject
* Patients who were taking or had been treated with Byetta® (exenatide) or other Glucagon-Like Peptide-1 agonists within 3 months before screening:
* Patients who were pregnant or breastfeeding
* Women of childbearing potential not protected by a highly effective contraceptive method of birth control (as defined for contraception in the Informed Consent Form and /or in a local protocol addendum) and/or who were unwilling or unable to be tested for pregnancy
* Patients with impaired renal function as shown by serum creatinine ≥1.5 mg/dL for males or ≥1.4 mg/dL for females at screening
* Patients with clinical evidence of active liver disease, or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2.5 times the upper limit of the normal range (ULN)
* Patients unlikely to comply with the protocol requirements (eg, illiterate, uncooperative, unable to return for scheduled visits, unlikely to complete the study)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of patients started on October 26, 2010 and the study was completed on May 7, 2012. Patients were screened in 60 centers in the United States of America, of which 59 centers randomized patients.
Pre-assignment Details: A total 623 patients were screened of whom 405 insulin naïve patients were randomized for the crossover phase. The most common reason for non randomization was glycosylated hemoglobin (HbA1c) value out of range at the screening visit as defined per protocol.
Groups:
- Pen (Period 1) / Vial & Syringe (Period 2): Crossover phase: patients randomized to the sequence: Lantus SoloSTAR® pen in Period 1 and Lantus vial and syringe in Period 2.
- Vial &Syringe (Period 1) / Pen (Period 2): Crossover phase: patients randomized to the sequence: Lantus vial and syringe in Period 1 and Lantus SoloSTAR pen in Period 2.
- SoloSTAR® Pen: Re-randomization phase and the observational phase: patients randomized to Lantus SoloSTAR® pen.
- Vial and Syringe: Re-randomization phase and the observational phase: patients randomized to Lantus Vial and Syringe.
Period: 4-week Crossover Phase - Period 1
Arm/Group | Pen (Period 1) / Vial & Syringe (Period 2) | Vial &Syringe (Period 1) / Pen (Period 2) | SoloSTAR® Pen | Vial and Syringe
Started | 202 | 203 | 0 | 0
TREATED | 202 | 200 | 0 | 0
Completed | 199 | 194 | 0 | 0
Not Completed | 3 | 9 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 6 | 0 | 0
Period: 4-week Crossover Phase - Period 2
Arm/Group | Pen (Period 1) / Vial & Syringe (Period 2) | Vial &Syringe (Period 1) / Pen (Period 2) | SoloSTAR® Pen | Vial and Syringe
Started | 199 | 194 | 0 | 0
TREATED | 199 | 194 | 0 | 0
Completed | 195 (28 patients were not re-randomized to the second phase of the study) | 188 (22 patients were not re-randomized to the second phase of the study) | 0 | 0
Not Completed | 4 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 4 | 5 | 0 | 0
Period: 6-week Re-randomization Phase
Arm/Group | Pen (Period 1) / Vial & Syringe (Period 2) | Vial &Syringe (Period 1) / Pen (Period 2) | SoloSTAR® Pen | Vial and Syringe
Started | 0 | 0 | 166 | 167
TREATED | 0 | 0 | 165 | 165
Completed | 0 | 0 | 159 | 156 (3 patients did not enter the observational phase of the study)
Not Completed | 0 | 0 | 7 | 11
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 3 | 2
Not completed — completed in error | 0 | 0 | 0 | 1
Period: 30-week Observational Phase
Arm/Group | Pen (Period 1) / Vial & Syringe (Period 2) | Vial &Syringe (Period 1) / Pen (Period 2) | SoloSTAR® Pen | Vial and Syringe
Started | 0 | 0 | 159 | 153
TREATED | 0 | 0 | 159 | 153
Completed | 0 | 0 | 153 | 140
Not Completed | 0 | 0 | 6 | 13
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 7
Not completed — Physician Decision | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics provided for the population randomized for the first phase of the study: crossover phase.
Groups:
- Crossover Phase: Pen / Vial & Syringe: Patients randomized to the sequence: Lantus SoloSTAR pen in Period 1 and Lantus vial and syringe in Period 2 for the 4-week crossover phase.
- Crossover Phase: Vial & Syringe / Pen: Patients randomized to the sequence: Lantus vial and syringe in Period 1 and Lantus SoloSTAR pen in Period 2 for the 4-week crossover phase.
- Total: Total of all reporting groups
Arm/Group | Crossover Phase: Pen / Vial & Syringe | Crossover Phase: Vial & Syringe / Pen | Total
Number analyzed (Participants) | 202 | 203 | 405
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 153 | 146 | 299
  >=65 years | 49 | 57 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.1) | 58.1 (10.9) | 57.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 88 | 188
  Male | 102 | 115 | 217
Body Weight [Mean (Standard Deviation); unit: kg] | 103.80 (26.43) | 98.48 (20.75) | 101.13 (23.87)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.93 (7.87) | 33.73 (6.64) | 34.83 (7.35)

OUTCOME MEASURES:

1. Primary Outcome: Patient Overall Preference
Description: The patient preference was assessed in terms of the difference in scores obtained from the overall preference question 14d "Overall, what is your level of preference for each of the insulin delivery systems?"
  5 points scale: from 1=Not preferred to 5= Always preferred
Time Frame: At week 4 (end of crossover phase)
Population: The modified intent-to-treat (mITT) population for the Patient Preference Questionnaire analysis consisted of all randomized patients who received at least one dose of Lantus via both insulin delivery systems and completed the questionnaire at Week 4. This analysis included patients who answered question 14d.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- SoloSTAR® Pen: Patients using the SoloSTAR® Pen during the crossover phase either at period 1 or at period 2 depending on the sequence allocated by randomization.
- Vial and Syringe: Patients using the Vial and Syringe during the crossover phase either at period 1 or at period 2 depending on the sequence allocated by randomization.
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 388 | 388
units on a scale | 4.75 (4.75) [4.65 to 4.85] | 2.45 [2.35 to 2.56]
Statistical Analysis 1: Comparison: SoloSTAR® Pen vs Vial and Syringe; The hypothesis was to determine whether patients have higher preference score for Lantus® SoloSTAR® pen compared to Lantus® vial/syringe. Differences of patient preference score greater than 0.5 were considered clinically meaningful. The power for detecting a true difference of 0.5 considering a standard deviation from 1.6 to 2.5, assuming 130 evaluable patients per arm and a two-sided test at 0.05 significance level ranged from 89% to more than 99%; Test type: Superiority or Other; p < 0.0001, ANOVA; The last observation carried forward (LOCF) method was applied to impute missing Week 4 overall patient preference values for ANOVA analysis; Mean Difference (Net) = 2.3, 95% CI 2-sided [2.15 to 2.44]

2. Secondary Outcome: Patient Preference Composite Score
Description: The patient preference composite score was the sum of the scores of the 3 following individual preference questions from the Patient preference Questionnaire:
  * Question 14a: How strongly do you prefer each of these insulin delivery systems to control blood sugar?
  * Question 14b: If using insulin for the first time, how strongly would you prefer using each of these delivery systems to overcome reluctance to use insulin?
  * Question 14c: How strongly would you prefer each insulin delivery system for long-term use?
  Each individual question scored from 1 to 5. The lowest score 1 indicated 'Not Preferred' and the highest score 5 indicated 'Always Preferred'. Therefore the total range of the composite score was 3 to 15.
Time Frame: At week 4 (end of crossover phase)
Population: The modified intent-to-treat (mITT) population for the Patient Preference Questionnaire analysis consisted of all randomized patients who received at least one dose of Lantus via both insulin delivery systems and completed the questionnaire at Week 4. This analysis included patients who answered to the 3 questions 14a, 14b and 14c.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 384 | 384
units on a scale | 14.2 [13.88 to 14.44] | 7.49 [7.21 to 7.77]

3. Secondary Outcome: Healthcare Professional's (HCP) Recommendation
Description: The overall recommendation score was obtained from the question 20d of the Healthcare Professional Questionnaire: "Overall, how strongly would you recommend each of the insulin delivery systems for your patients?"
  5 points scale: from 1= Not Recommended to 5= Recommended
Time Frame: At week 4 (end of crossover phase)
Population: The HCP Questionnaire analysis population consisted of HCPs:
  * who treated at least 1 randomized patient during the crossover phase and this(these) patient(s) received at least one dose of Lantus via both insulin delivery systems during the crossover phase
  * who completed the HCP Questionnaire.
Measure: Median (Full Range); unit: units on a scale
Groups:
- SoloSTAR® Pen: SoloSTAR® Pen used during the crossover phase either at period 1 or at period 2
- Vial and Syringe: Vial and Syringe used during the crossover phase either at period 1 or at period 2
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 135 | 135
units on a scale | 5.0 [4 to 5] | 3.0 [1 to 5]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Time Frame: From week 4 (baseline for re-randomization phase) to week 10 (end of re-randomization phase)
Population: The mITT population for Re-randomization and Observational Phases consisted of all patients who were re-randomized, received at least one dose of Lantus after re-randomization, and had both a re-randomization baseline assessment and at least one post re-randomization assessment of FPG measured during the on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- SoloSTAR® Pen: Patients randomized to SoloSTAR® Pen during the Re-randomization period (Week 4 to Week 10)
- Vial and Syringe: Patients randomized to Vial and Syringe during the Re-randomization period (Week 4 to Week 10)
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 154 | 150
mg/dL | -14.3 (2.87) | -14.5 (2.91)

5. Secondary Outcome: Percentage of Patients Achieving Fasting Plasma Glucose (FPG) <110 mg/dL
Time Frame: At week 10 (end of re-randomization phase)
Population: The mITT population for Re-randomization and Observational Phases consisted of all patients who were re-randomized, received at least one dose of Lantus after re-randomization, and had a re-randomization baseline assessment FPG > or = 110 (week 4) and at least one post re-randomization assessment of FPG.
Measure: Number; unit: percentage of patients
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 125 | 128
percentage of patients | 28.8 | 30.5

6. Secondary Outcome: Change in Lantus Dose Injected Per Day
Time Frame: From week 4 (baseline for re-randomization phase) to week 10 (end of re-randomization phase)
Population: The mITT population for Re-randomization and Observational Phases consisted of all patients who were re-randomized, received at least one dose of Lantus after re-randomization, and had both a re-randomization baseline assessment and at least one post re-randomization assessment of FPG.
Measure: Least Squares Mean (Standard Error); unit: U (insulin unit)
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 159 | 155
U (insulin unit) | 6.361 (0.786) | 6.336 (0.796)

7. Secondary Outcome: Percentage of Patients Achieving HbA1c Goal
Description: Percentage of patients achieving HbA1c < 7% at Week 40 (end of the observational phase)
Time Frame: measured at week 40 or at study discontinuation
Population: Patients from the mITT population for Re-randomization and Observational Phases who had at least one post re-randomization assessment of HbA1c.
Measure: Number; unit: percentage of patients
Groups:
- SoloSTAR® Pen: Patients randomized to SoloSTAR® Pen during the Re-randomization phase (from Week 4 to Week 10) and the Observational phase (from Week 10 to Week 40).
- Vial and Syringe: Patients randomized to Vial and Syringe during the Re-randomization phase (from Week 4 to Week 10) and the Observational phase (from Week 10 to Week 40).
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 159 | 154
percentage of patients | 37.7 | 37.0

8. Secondary Outcome: Time to First Observation of HbA1c <7%
Time Frame: From week 10 to week 40 (observational phase)
Population: The mITT population for Re-randomization and Observational Phases consisted of all patients who were re-randomized, received at least one dose of Lantus after re-randomization, and had both a re-randomization baseline assessment and at least one post re-randomization assessment of HbA1c.
Measure: Median (95% Confidence Interval); unit: Days since Re-randomization (week 4)
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 155 | 149
Days since Re-randomization (week 4) | 166 [88 to 248] | 168 [91 to 250]

9. Secondary Outcome: Percentage of Patients Who Discontinued Investigational Product (IP) During the Crossover Phase
Time Frame: From baseline to week 4 (crossover phase)
Population: Randomized population (crossover phase) exposed to at least one dose of the IP
Measure: Number; unit: percentage of patients
Groups:
- SoloSTAR® Pen (Period 1): Patients using SoloSTAR® pen during period 1 of the crossover phase.
- Vial and Syringe (Period 2): Patients using Vial and Syringe during period 2 of the crossover phase.
- SoloSTAR® Pen (Period 2): Patients using SoloSTAR® pen during period 2 of the crossover phase.
- Vial and Syringe (Period 1): Patients using Vial and Syringe during period 1 of the crossover phase.
Arm/Group | SoloSTAR® Pen (Period 1) | Vial and Syringe (Period 2) | SoloSTAR® Pen (Period 2) | Vial and Syringe (Period 1)
Number analyzed (Participants) | 202 | 199 | 194 | 200
percentage of patients | 1.49 | 2.01 | 3.09 | 3.00

10. Secondary Outcome: Percentage of Patients Who Discontinued Investigational Product During the Re-randomization Phase
Time Frame: From week 4 to week 10 (re-randomization phase)
Population: Re-randomized population at week 4 exposed to at least one dose of the IP
Measure: Number; unit: percentage of patients
Groups:
- SoloSTAR® Pen: Patients using SoloSTAR® pen during the re-randomization phase.
- Vial and Syringe: Patients using Vial and Syringe during the re-randomization phase.
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 165 | 165
percentage of patients | 3.6 | 5.5

11. Secondary Outcome: Percentage of Patients Who Discontinued Investigational Product During the Observational Phase
Time Frame: From week 10 to week 40 (observational phase)
Population: Re-randomized population at week 4 and included in the observational phase at week 10 and exposed to at least one dose of the IP
Measure: Number; unit: percentage of patients
Groups:
- SoloSTAR® Pen: Patients using SoloSTAR® pen during the observational phase.
- Vial and Syringe: Patients using Vial and Syringe during the observational phase.
Arm/Group | SoloSTAR® Pen | Vial and Syringe
Number analyzed (Participants) | 159 | 153
percentage of patients | 3.8 | 8.5

12. Other Pre Specified Outcome: Number of Patients With Hypoglycemic Events
Description: The hypoglycemic event was to be recorded on the electronic case report form hypoglycemia page and had to fit in one of the following categories: Mild-to-moderate hypoglycemia (36 mg/dL ≤ Self Monitored Blood Glucose (SMBG) <70mg/dL), Severe hypoglycemia (assistance of another person is required, and either a recorded SMBG <36 mg/dL, or treatment with oral carbohydrates, intravenous glucose or glucagon with prompt response) or Hypoglycemia symptoms with or without SMBG values with a documented SMBG >70 mg/dL, or no recorded SMBG value. Only hypoglycemia events associated with coma, loss of consciousness or seizure were considered serious adverse event (SAEs).
Time Frame: each study phase (crossover, re-randomization, observational) up to 40 weeks
Population: The safety population for each phase (crossover, re-randomization, observational) was the total treated population defined as all the patients who were randomized and exposed to at least one dose of Lantus during that phase.
Measure: Number; unit: participants having reported the event
Groups:
- Crossover Phase: SoloSTAR® Pen: Patients using the SoloSTAR® Pen during the crossover phase either at period 1 or at period 2 depending on the sequence allocated by randomization.
- Crossover Phase: Vial and Syringe: Patients using Vial and Syringe during the crossover phase either at period 1 or at period 2 depending on the sequence allocated by randomization.
- Re-randomization Phase: SoloSTAR® Pen: Patients randomized to SoloSTAR® Pen during the Re-randomization period (Week 4 to Week 10)
- Re-randomization Phase: Vial and Syringe: Patients randomized to Vial and Syringe during the Re-randomization period (Week 4 to Week 10)
- Observational Phase: SoloSTAR® Pen: Patients using SoloSTAR® Pen during the Observational phase (from Week 10 to Week 40)
- Observational Phase: Vial and Syringe: Patients using Vial and Syringe during the Observational phase (from Week 10 to Week 40)
Arm/Group | Crossover Phase: SoloSTAR® Pen | Crossover Phase: Vial and Syringe | Re-randomization Phase: SoloSTAR® Pen | Re-randomization Phase: Vial and Syringe | Observational Phase: SoloSTAR® Pen | Observational Phase: Vial and Syringe
Number analyzed (Participants) | 396 | 399 | 165 | 165 | 159 | 153
participants having reported the event
  Hypoglycemic event with or without SMBG | 72 | 83 | 43 | 48 | 76 | 73
  Hypoglycemia with SMBG | 69 | 81 | 38 | 47 | 75 | 71
  Symptomatic hypoglycemia | 57 | 68 | 37 | 37 | 61 | 61
  Hypoglycemia, assistance required | 3 | 2 | 2 | 5 | 8 | 11
  Severe hypoglycemia | 3 | 2 | 2 | 4 | 7 | 11
  Serious hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The median of exposure to each device was 14 days during the crossover phase. The median of exposure was 43 days in both arms during the re-randomization phase. During the observational phase, it was 209 days in the pen arm and 210 days in the vial arm.
Arm/Group | Crossover Phase: SoloSTAR® Pen | Crossover Phase: Vial and Syringe | Re-randomization Phase: SoloSTAR® Pen | Re-randomization Phase: Vial and Syringe | Observational Phase: SoloSTAR® Pen | Observational Phase: Vial and Syringe
Serious Adverse Events (participants affected / at risk) | 4/396 | 1/399 | 1/165 | 0/165 | 16/159 | 14/153
Other Adverse Events (participants affected / at risk) | 18/396 | 5/399 | 12/165 | 14/165 | 35/159 | 34/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Phase: SoloSTAR® Pen (N=396) | Crossover Phase: Vial and Syringe (N=399) | Re-randomization Phase: SoloSTAR® Pen (N=165) | Re-randomization Phase: Vial and Syringe (N=165) | Observational Phase: SoloSTAR® Pen (N=159) | Observational Phase: Vial and Syringe (N=153)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cauda equina syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Colon neoplasm (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Osteomyelitis (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pancreatic mass (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural complication (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1 | 0
Transurethral bladder resection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Urethral obstruction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Phase: SoloSTAR® Pen (N=396) | Crossover Phase: Vial and Syringe (N=399) | Re-randomization Phase: SoloSTAR® Pen (N=165) | Re-randomization Phase: Vial and Syringe (N=165) | Observational Phase: SoloSTAR® Pen (N=159) | Observational Phase: Vial and Syringe (N=153)
Nasopharyngitis (Infections and infestations) | 5 | 0 | 6 | 4 | 7 | 13
Sinusitis (Infections and infestations) | 4 | 1 | 2 | 6 | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 4 | 1 | 14 | 12
Oedema peripheral (General disorders) | 2 | 2 | 0 | 3 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.